CLINICAL TRIAL: NCT06312631
Title: Benefits of a Home Grip Assistance Glove on the Use of the Upper Limb and Compliance Factors in Brain-injured Adults: Comparative Multicenter Study
Brief Title: Home Grip Assistance Glove on the Use of the Upper Limb and Compliance Factors in Brain-injured Adults
Acronym: ECO-HAND-AVC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: RC31/21/0342
Record Dates: First submitted 2024-03-08; First posted 2024-03-15 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Stroke
Keywords: brain-injured adult
MeSH Terms: conditions — Stroke | interventions — Surveys and Questionnaires; Self-Help Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (8):
- Task handover model #1 (Experimental): At each visit, the patient will perform the tasks with the gripping glove (A) or without the gripping glove (B).
  The order of administration "with then without the glove (AB)" or "without then with the glove (BA)" is drawn at random for each patient.
  The 1st model follows the following diagram:
  Visit T1 = AB; Visit T2 = AB; Visit T3 = AB
  Interventions: Device: Putting on the gripping glove; Other: ULPA questionnaire; Other: Motor Activity Log (MAL) Questionnaire; Other: Fugl-Meyer Assessment Upper Extremity (FMA-UE) questionnaire; Other: Score Action Arm Research Test; Other: EuroQol five-level (EQ-5D-5L) questionnaire; Other: Quebec User Evaluation of Satisfaction with Assistive Technology; Other: Psychosocial Impact of Assistive Devices Scale (PIADS); Other: Goal Attainment Scale (GAS); Other: installation and collection of accelerometers
- Task handover model #2 (Experimental): At each visit, the patient will perform the tasks with the gripping glove (A) or without the gripping glove (B).
  The order of administration "with then without the glove (AB)" or "without then with the glove (BA)" is drawn at random for each patient.
  The 2nd model follows the following diagram:
  Visit T1 = BA ; Visit T2 = AB ; Visit T3 = AB
  Interventions: Device: Putting on the gripping glove; Other: ULPA questionnaire; Other: Motor Activity Log (MAL) Questionnaire; Other: Fugl-Meyer Assessment Upper Extremity (FMA-UE) questionnaire; Other: Score Action Arm Research Test; Other: EuroQol five-level (EQ-5D-5L) questionnaire; Other: Quebec User Evaluation of Satisfaction with Assistive Technology; Other: Psychosocial Impact of Assistive Devices Scale (PIADS); Other: Goal Attainment Scale (GAS); Other: installation and collection of accelerometers
- Task handover model #3 (Experimental): At each visit, the patient will perform the tasks with the gripping glove (A) or without the gripping glove (B).
  The order of administration "with then without the glove (AB)" or "without then with the glove (BA)" is drawn at random for each patient.
  The 3rd model follows the following diagram:
  Visit T1 = AB ; Visit T2 = BA ; Visit T3 = AB
  Interventions: Device: Putting on the gripping glove; Other: ULPA questionnaire; Other: Motor Activity Log (MAL) Questionnaire; Other: Fugl-Meyer Assessment Upper Extremity (FMA-UE) questionnaire; Other: Score Action Arm Research Test; Other: EuroQol five-level (EQ-5D-5L) questionnaire; Other: Quebec User Evaluation of Satisfaction with Assistive Technology; Other: Psychosocial Impact of Assistive Devices Scale (PIADS); Other: Goal Attainment Scale (GAS); Other: installation and collection of accelerometers
- Task handover model #4 (Experimental): At each visit, the patient will perform the tasks with the gripping glove (A) or without the gripping glove (B).
  The order of administration "with then without the glove (AB)" or "without then with the glove (BA)" is drawn at random for each patient.
  The 4th model follows the following diagram:
  Visit T1 = AB ; Visit T2 = AB ; Visit T3 = BA
  Interventions: Device: Putting on the gripping glove; Other: ULPA questionnaire; Other: Motor Activity Log (MAL) Questionnaire; Other: Fugl-Meyer Assessment Upper Extremity (FMA-UE) questionnaire; Other: Score Action Arm Research Test; Other: EuroQol five-level (EQ-5D-5L) questionnaire; Other: Quebec User Evaluation of Satisfaction with Assistive Technology; Other: Psychosocial Impact of Assistive Devices Scale (PIADS); Other: Goal Attainment Scale (GAS); Other: installation and collection of accelerometers
- Task handover model #5 (Experimental): At each visit, the patient will perform the tasks with the gripping glove (A) or without the gripping glove (B).
  The order of administration "with then without the glove (AB)" or "without then with the glove (BA)" is drawn at random for each patient.
  The 5th model follows the following diagram:
  Visit T1 = BA ; Visit T2 = BA ; Visit T3 = AB
  Interventions: Device: Putting on the gripping glove; Other: ULPA questionnaire; Other: Motor Activity Log (MAL) Questionnaire; Other: Fugl-Meyer Assessment Upper Extremity (FMA-UE) questionnaire; Other: Score Action Arm Research Test; Other: EuroQol five-level (EQ-5D-5L) questionnaire; Other: Quebec User Evaluation of Satisfaction with Assistive Technology; Other: Psychosocial Impact of Assistive Devices Scale (PIADS); Other: Goal Attainment Scale (GAS); Other: installation and collection of accelerometers
- Task handover model #6 (Experimental): At each visit, the patient will perform the tasks with the gripping glove (A) or without the gripping glove (B).
  The order of administration "with then without the glove (AB)" or "without then with the glove (BA)" is drawn at random for each patient.
  The 6th model follows the following diagram:
  Visit T1 = BA ; Visit T2 = AB ; Visit T3 = BA
  Interventions: Device: Putting on the gripping glove; Other: ULPA questionnaire; Other: Motor Activity Log (MAL) Questionnaire; Other: Fugl-Meyer Assessment Upper Extremity (FMA-UE) questionnaire; Other: Score Action Arm Research Test; Other: EuroQol five-level (EQ-5D-5L) questionnaire; Other: Quebec User Evaluation of Satisfaction with Assistive Technology; Other: Psychosocial Impact of Assistive Devices Scale (PIADS); Other: Goal Attainment Scale (GAS); Other: installation and collection of accelerometers
- Task handover model #7 (Experimental): At each visit, the patient will perform the tasks with the gripping glove (A) or without the gripping glove (B).
  The order of administration "with then without the glove (AB)" or "without then with the glove (BA)" is drawn at random for each patient.
  The 7th model follows the following diagram:
  Visit T1 = AB ; Visit T2 = BA ; Visit T3 = BA
  Interventions: Device: Putting on the gripping glove; Other: ULPA questionnaire; Other: Motor Activity Log (MAL) Questionnaire; Other: Fugl-Meyer Assessment Upper Extremity (FMA-UE) questionnaire; Other: Score Action Arm Research Test; Other: EuroQol five-level (EQ-5D-5L) questionnaire; Other: Quebec User Evaluation of Satisfaction with Assistive Technology; Other: Psychosocial Impact of Assistive Devices Scale (PIADS); Other: Goal Attainment Scale (GAS); Other: installation and collection of accelerometers
- Task handover model #8 (Experimental): At each visit, the patient will perform the tasks with the gripping glove (A) or without the gripping glove (B).
  The order of administration "with then without the glove (AB)" or "without then with the glove (BA)" is drawn at random for each patient.
  The 8th model follows the following diagram:
  Visit T1 = BA ; Visit T2 = BA ; Visit T3 = BA
  Interventions: Device: Putting on the gripping glove; Other: ULPA questionnaire; Other: Motor Activity Log (MAL) Questionnaire; Other: Fugl-Meyer Assessment Upper Extremity (FMA-UE) questionnaire; Other: Score Action Arm Research Test; Other: EuroQol five-level (EQ-5D-5L) questionnaire; Other: Quebec User Evaluation of Satisfaction with Assistive Technology; Other: Psychosocial Impact of Assistive Devices Scale (PIADS); Other: Goal Attainment Scale (GAS); Other: installation and collection of accelerometers

INTERVENTIONS:
Device: Putting on the gripping glove — taking measurements and putting the gripping glove on the patient
Other: ULPA questionnaire — The evaluation of the effectiveness of the gripping glove on the performance of the upper limb in daily life will be evaluated using the ULPA score.
  The investigator asks the patient to perform a task and the ULPA collects the total number of errors made by the patient (inability/omission, imprecision, repetition, time to complete the task)
Other: Motor Activity Log (MAL) Questionnaire — The MAL is a self-assessment of the integration of the upper limb into daily life. This measurement allows a quantified evaluation of the perceived performance of the use of the upper limb in the actions of daily life.
  The patient will answer 30 questions about daily life and for each item, rate the quantity from 0 to 5: 0 = never uses the hemiplegic arm and 5 = uses as much as before the accident
Other: Fugl-Meyer Assessment Upper Extremity (FMA-UE) questionnaire — This questionnaire assesses the motor selectivity of the upper limb. Several questions are asked about the movements that the patient can perform and to each question, the patient can answer either 0 (minimum) and 2 (maximum).
Other: Score Action Arm Research Test — This questionnaire evaluates 4 different actions: Grasping an object (6 different objects to grasp), holding an object (4 different objects), pinching an object (6 different objects) and the overall movements made by the patient (3 different overall movements).
  For each item, each object or each movement evaluated, the patient must rate the task on a scale of 0 to 3 (0=cannot perform any part of the test and 3=performs the test normally)
Other: EuroQol five-level (EQ-5D-5L) questionnaire — This questionnaire assesses the patient's state of health. 5 items are proposed (mobility, autonomy, current activity, pain, anxiety) and for each the patient must check one of the 5 propositions (no problem, mild problems, moderate problems, severe problems, incapable). The patient must also rate their state of health on a scale of 0 to 100.
Other: Quebec User Evaluation of Satisfaction with Assistive Technology — This questionnaire assesses satisfaction with the technical aid (here the gripping glove) and the related services. The technique and related services will be evaluated by items provided to the patient and he will have to rate for each of them a score between 1 and 5 (1 = not satisfied at all and 5 = very satisfied)
Other: Psychosocial Impact of Assistive Devices Scale (PIADS) — This questionnaire measures the effect of technical aids on the psychosocial level. 26 sentences or words are offered to the patient concerning his psychological state and the patient must evaluate them between -3 and 3 (-3 = decreased and +3: increased)
Other: Goal Attainment Scale (GAS) — Carrying out an activity in the patient's real context is assessed using the Goal Attainment Scale (GAS). The doctor gives the patient objectives to achieve and the patient must give the quotation for each objective between initial state (-2), expected result (0) and best possible result (2)
Other: installation and collection of accelerometers — The accelerometer quantitatively reports the spontaneous use of the upper limb in daily life. It counts the number of voluntary movements of the upper limbs. The amount of movement of the paretic upper limb will be expressed as a percentage of the movements of the non-paretic limb.

SUMMARY:
On a functional level, performing the actions of daily life requires coordinated activity of the muscles of the upper limbs. The quality of motor recovery and/or technical assistance aimed at compensating for the movement deficit of the paretic upper limb (MSP) determines the possibilities of using the upper limb (MS) in activities of daily life.

Interventions in the chronic phase of stroke aim to return home. The integration of the paretic upper limb into daily life activities is a major issue regarding the prognosis of recovery of use of the upper limb. Independence in daily life becomes an ultimate goal to take charge of.

This study focuses on a new technical aid device, standard orthosis type, expanding the range of gripping gloves: the SaeboGlove in everyday environments. These MS orthoses help improve the use and function of the MSP in post-stroke adults as well as their independence and participation in society.

ELIGIBILITY:
Inclusion Criteria:

* Patient suffering from a motor deficit of the upper limb resulting from an ischemic or hemorrhagic stroke, hemispheric or brainstem, confirmed by brain imaging ;
* Patient who suffered a stroke more than three months ago;
* Patient unable to actively extend long fingers (hand opening) to voluntarily grasp an empty glass (upper and lower diameter of 7 and 6 cm respectively, height of 12 to 15 cm, weight of 125g, identical to equipment used for ARAT), with a palmar grip (cylindrical grip), while the subject can hold the previously placed glass passively in the hand;
* Patient capable of passively opening the hand sufficient to grasp the glass when the gripping glove is put on, with the possibility of actively closing the hand;
* Patient with the ability to put on and remove the SaeboGlove® gripping glove with the help of a third person if necessary and/or available.
* Patient with a smartphone, tablet and/or computer compatible with video taking and teleconsultation.
* Free, informed and signed consent by the participant and/or the person having guardianship and the investigator (at the latest on the day of inclusion and before any examination required by the research);
* Person affiliated to or beneficiary of a social security system.

Exclusion Criteria:

* Patient presenting retraction or stiffness of the fingers and wrist preventing complete extension of the long fingers and thumb, the wrist being at 15° extension;
* Patient with moderate or severe muscular spasticity of the wrist flexors and the long and short flexors of the fingers and thumb (Modified Ashworth Scale ≥ 3);
* Patient with limited active elbow extension, not allowing the ipsilateral knee to be reached with the hand, the subject being seated with the trunk vertical (approach limitation);
* Patient with an active anterior shoulder elevation range of less than 15°;
* Patient with other upper limb deficiencies likely to influence participation;
* Patient and/or entourage who do not have access to teleconsultation, and/or can be reached remotely;
* Patient with severe aphasia, Boston Diagnostic Aphasia Examination (BDAE) ≤ 3;
* Presence of moderate or severe edema localized to the wrist and hand;
* Patient allergic to Latex
* History of upper limb surgery less than 6 months old.
* Pregnant and/or breastfeeding women
* Patient deprived of liberty (detained/incarcerated);
* Patient under judicial protection
* Impossibility of giving the person informed information and ensuring the subject's compliance due to impaired physical and/or psychological health

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-03-26 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the effectiveness of the gripping glove | 6 months
  The evaluation of the effectiveness of the gripping glove on the performance of the upper limb in daily life will be evaluated using the ULPA score and compared between the 2 conditions (with and without the glove) in the performance of a daily activity.

SECONDARY OUTCOMES:
Evaluation of the performance of an activity in the real context of the patient | 6 months
  The performance of an activity in the real context of the patient will be evaluated using the GAS. Information is collected from the person and/or their entourage at each visit, assessed during visits T1 (14 days), T2 (3 months) and T3 (6 months) by the assessor (occupational therapist) from each center.
Evaluation of factual spontaneous use of the upper limb in daily life | 6 months
  Factual spontaneous use of the upper limb in daily life will be measured using a wrist accelerometer. The movement will be compared between T0, T2 (3 months) and T3 (6 months).
Evaluation of the perceived performance of the use of the paretic upper limb | 6 months
  The perceived performance of the use of the paretic upper limb will be evaluated using the MAL at T0, T2 (3 months) and T3 (6 months).
Assessment of the quality of voluntary motor skills of the upper limb | 6 months
  The quality of voluntary motor skills of the upper limb will be assessed with the FMA at T0, T2 (3 months) and T3 (6 months), without wearing the gripping glove.
Assessment of gripping abilities | 6 months
  Grasping abilities will be assessed by the ARAT at T0, T2 (3 months) and T3 (6 months), without wearing the gripping glove.
Quality of life assessment | 6 months
  Quality of life, assessed using the EQ-5D-5L, will be explored at T0, T2 (3 months) and T3 (6 months).
Evaluation of satisfaction and tolerance | 6 months
  Satisfaction and tolerance will be assessed by the patient with the QUEST version 2.0 questionnaire, at the end of the T3 visit (6 months).
Evaluation of the psycho-social impact | 6 months
  The psycho-social impact will be assessed with the F-PIADS questionnaire during visits to T2 (3 months) T3 (6 months), by the evaluator (occupational therapist) from each center.

CONTACTS AND LOCATIONS:
Overall Officials: Claire VILLEPINTE, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Claire VILLEPINTE, Toulouse, France

IPD SHARING:
Plan to Share IPD: No